CLINICAL TRIAL: NCT00971048
Title: Evaluation of the Effects of HP828-101 Versus Standard of Care in the Management of Partial or Full Thickness Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 828-101-09-013
Record Dates: First submitted 2009-08-27; First posted 2009-09-03 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Foot Ulcers; Pressure Ulcers
Keywords: pressure ulcers; PU; diabetic foot ulcers; DFU; Bates-Jensen Wound Assessment
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HP828-101 (Experimental)
  Interventions: Device: HP828-101
- Standard of Care (Active Comparator): For DFU SoC is a hydrogel. For PU SoC is a hydrocolloid gel.
  Interventions: Device: Hydrogel/Hydrocolloid

INTERVENTIONS:
Device: HP828-101 — Topical test article applied once daily
  Other Names: New device, no brand name identified-Code name is HP828-101
  Arms: HP828-101
Device: Hydrogel/Hydrocolloid — Hydrogel for DFU and Hydrocolloid for PU (3M Tegaderm Hydrogel for DFU; ConvaTec DuoDERM Hydroactive Gel for PU); Topical test articles applied once daily
  Other Names: 3M Tegaderm Hydrogel for DFU; ConvaTec DuoDERM Hydroactive Gel for PU
  Arms: Standard of Care

SUMMARY:
To compare HP828-101 to standard of care for the management of partial or full thickness wounds

DETAILED DESCRIPTION:
The primary objective is to compare HP828-101 to standard of care for the management of partial or full thickness wounds, evaluated using the Bates Jensen Wound Assessment Tool (BWAT).

The secondary objectives are comparison of the proportion of subjects with wound closure by day 22, comparison of pain assessed using a visual analog scale (VAS), and evaluation of moist wound environment as per the BWAT.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent document must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams. In addition, the informed consent document must be signed and dated by the individual who consents the subject before conducting Visit 1. A photocopy of the signed informed consent document must be provided to the subject, and the original signed document placed in the subject's chart. For subjects that agree to have their wound photographed for the trial, a photo release consent form must be signed and documented as well.
* Age 18 years or older, of either sex, and of any race or skin type, provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* Females, if of child-bearing potential, have a negative urine pregnancy test and agree to use acceptable contraception during the study. Adequate birth control methods are defined as: hormonal-topical, oral, implantable, or injectable contraceptives; mechanical-spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or surgical sterilization of partner.
* Have a partial or full thickness PU on the foot or ankle or DFU of <= 6 months duration and between ≥1.0 and ≤ 12.0 cm² in area.
* Are willing to make all required study visits.
* Are willing to follow instructions, in the opinion of the Investigator.
* Have, within 12 weeks prior to randomization, a serum albumin level ≥ 2.0 g/dL (20 g/L); Alkaline phosphatase, AST, ALT, serum creatinine, and BUN levels < 3 x upper limit of normal; HbA1C ≤ 12%; and Hemoglobin >= 8 g/dL. The most recently obtained value must be evaluated against these criteria. Please refer to Appendix 18.1.5
* Have arterial supply adequacy confirmed by an Ankle Brachial Index (ABI) >= 0.7 and ≤ 1.1 or if the ABI is > 1.1, either a TcPO2 >= 40 mmHg, as measured on the foot, or great toe pressure ≥ 50 mm/Hg,
* For ulcers that will require surgical debridement prior to enrollment, the wound must be expected to remain a partial thickness wound after debridement.

Exclusion Criteria:

* Have a known hypersensitivity to any of the test articles or their components.
* Have received therapy with another investigational agent within thirty (30) days of Visit 1.
* Are pregnant or nursing.
* Have clinical evidence of bacterial or fungal infection of the wound per visual/clinical assessment.
* Have a severe burn, immunodeficiency disorder, hematologic disorder, or metastatic malignancy.
* Have had documented osteomyelitis on the target ulcer leg within 6 months preceding the screening visit.
* Have severe edema of the target ulcer leg.
* If being treated with Xenaderm, must stop treatment prior to enrolling in the study.
* Have received treatment with glucocorticoids for > 10 consecutive days within 6 months prior to the start of the study.
* Have received chemotherapy or radiation therapy within the past 5 years.
* Therapy of the target ulcer with tissue-engineered cell-based skin equivalents within 30 days preceding the Screening Visit (e.g., Apligraf®).
* Therapy of the target ulcer with topical growth factors within 1 week preceding the Screening Visit.
* Current therapy with systemic or topical antibiotics or systemic therapy with cytotoxic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Innes Cargill, PhD, Study Director — Healthpoint, Ltd
Locations (11):
- United States (11):
  - Trovare Clinical Research, Bakersfield, California
  - Absolute Foot Care, Chula Vista, California
  - Roy Kroeker, Fresno, California
  - Innovative Medical Technologies, Los Angeles, California
  - San Diego Research Center, San Diego, California
  - Foot and Ankle Associates of Florida, Altamonte Springs, Florida
  - Weil Foot and Ankle Institute, Des Plaines, Illinois
  - Prigoff-Bowers LLP, Dallas, Texas
  - Richard Galperin, DPM, Dallas, Texas
  - Robert Wunderlich, DPM, San Antonio, Texas
  - Dixie Regional Wound Clinic, St. George, Utah

REFERENCES:
- [Background] Ovington LG. The evolution of wound management: ancient origins and advances of the past 20 years. Home Healthc Nurse. 2002 Oct;20(10):652-6. doi: 10.1097/00004045-200210000-00009. PMID 12394337
- [Background] Winter GD. Formation of the scab and the rate of epithelisation of superficial wounds in the skin of the young domestic pig. 1962. J Wound Care. 1995 Sep;4(8):366-7; discussion 368-71. No abstract available. PMID 7553187
- [Background] HINMAN CD, MAIBACH H. EFFECT OF AIR EXPOSURE AND OCCLUSION ON EXPERIMENTAL HUMAN SKIN WOUNDS. Nature. 1963 Oct 26;200:377-8. doi: 10.1038/200377a0. No abstract available. PMID 14087904
- [Background] Andersen CA, Roukis TS. The diabetic foot. Surg Clin North Am. 2007 Oct;87(5):1149-77, x. doi: 10.1016/j.suc.2007.08.001. PMID 17936480
- [Background] Frykberg RG. Epidemiology of the diabetic foot: ulcerations and amputations. Adv Wound Care. 1999 Apr;12(3):139-41. No abstract available. PMID 10655794
- [Background] Sussman C, Bates-Jensen B. Wound Care - A Collaborative Practice Manual for Health Professionals. 3rd Ed. Philadelphia: Lippincott Williams & Wilkins, 2006.
- [Background] Hess CT. Wound Care. 5th Ed ed. Philadelphia: Lippincott Williams & Wilkins, 2005.
- [Background] Steed DL, Attinger C, Colaizzi T, Crossland M, Franz M, Harkless L, Johnson A, Moosa H, Robson M, Serena T, Sheehan P, Veves A, Wiersma-Bryant L. Guidelines for the treatment of diabetic ulcers. Wound Repair Regen. 2006 Nov-Dec;14(6):680-92. doi: 10.1111/j.1524-475X.2006.00176.x. No abstract available. PMID 17199833
- [Background] Agren MS. An amorphous hydrogel enhances epithelialisation of wounds. Acta Derm Venereol. 1998 Mar;78(2):119-22. doi: 10.1080/000155598433449. PMID 9534889
- [Background] Whitney J, Phillips L, Aslam R, Barbul A, Gottrup F, Gould L, Robson MC, Rodeheaver G, Thomas D, Stotts N. Guidelines for the treatment of pressure ulcers. Wound Repair Regen. 2006 Nov-Dec;14(6):663-79. doi: 10.1111/j.1524-475X.2006.00175.x. No abstract available. PMID 17199832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults 18 years of age and older who had a DFU or PU on the foot that was a partial or full thickness wound
Groups:
- HP828-101 Treating DFU: HP828-101 : Topical test article approximately the size of a nickel, applied once daily Treatment group had diabetic foot ulcers (DFU)
- Standard of Care Treating DFU: For diabetic foot ulcers (DFU) Standard of Care (SoC) is a hydrogel
  Hydrogel for DFU (3M Tegaderm Hydrogel)
- HP828-101 Treating PU: HP828-101 : Topical test article approximately the size of a nickel, applied once daily Treatment group had pressure ulcers (PU)
- Standard of Care Treating PU: For Pressure Ulcers (PU) Standard of Care (SoC) was a hydrocolloid gel
  Hydrocolloid for PU: Topical test articles applied once daily (ConvaTec DuoDERM Hydroactive Gel for PU)
Period: Overall Study
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU
Started | 30 | 33 | 12 | 13
Completed | 29 | 31 | 11 | 11
Not Completed | 1 | 2 | 1 | 2
Not completed — Protocol Violation | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- HP828-101 Treating DFU: HP828-101 : Topical test article applied once daily Treatment group had diabetic foot ulcers (DFU)
- Standard of Care Treating DFU: For diabetic foot ulcers (DFU) Standard of Care (SoC) is a hydrogel
  Hydrogel for DFU(3M Tegaderm Hydrogel)
- HP828-101 Treating PU: HP828-101 : Topical test article applied once daily Treatment group had pressure ulcers (PU)
- Total: Total of all reporting groups
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU | Total
Number analyzed (Participants) | 30 | 33 | 12 | 13 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 7 | 7 | 49
  >=65 years | 12 | 16 | 5 | 6 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (13.5) | 63.5 (10.4) | 61.3 (12.6) | 64.1 (17.0) | 62.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 4 | 5 | 30
  Male | 19 | 23 | 8 | 8 | 58
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 12 | 13 | 88

OUTCOME MEASURES:

1. Primary Outcome: Adequate Management of the Wound Assessed by a Left Movement (Improvement) in the Modified Bates Jensen Wound Assessment Tool.
Description: Modified Bates-Jensen Wound Assessment (BWAT-m) Scores for those characteristics measured (wound size, depth, edges, undermining, necrotic tissue type and amount, exudate type and amount, periwound color and edema, granulation tissue, and epithelialization) were each graded on a 5-point scale, with 1 being the best and 5 being the worst.
Time Frame: 22 - 29 days
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU
Number analyzed (Participants) | 30 | 33 | 12 | 13
units on a scale
  Day 22 | 20.28 (0.89) | 21.38 (0.85) | 20.94 (1.63) | 20.59 (1.57)
  Day 29 | 20.12 (0.98) | 18.71 (0.93) | 19.78 (1.67) | 17.28 (1.61)

2. Secondary Outcome: Number of Participants With Wound Closure by Day 22.
Time Frame: 22 days
Measure: Number; unit: Subjects
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU
Number analyzed (Participants) | 30 | 33 | 12 | 13
Subjects | 5 | 1 | 1 | 3

3. Secondary Outcome: Pain Assessed by a 100-mm VAS Scale.
Description: 100-mm VAS scale was used to evaluate pain, with 1 being healthy tissue (no pain) up to 100 (wound degeneration and severe pain)
Time Frame: At every visit: Day 8, Day 15, Day 22, Day 29
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: VAS Pain Scores
Groups:
- HP828-101 Treating DFU: HP828-101 : Topical test article applied approximately the size of a nickel, once daily Treatment group had diabetic foot ulcers (DFU)
- HP828-101 Treating PU: HP828-101 : Topical test article applied approximately the size of a nickel, once daily Treatment group had pressure ulcers (PU)
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU
Number analyzed (Participants) | 30 | 33 | 12 | 13
VAS Pain Scores
  Day 8 | 8.92 (1.84) | 4.85 (1.75) | 4.76 (1.21) | 6.99 (1.16)
  Day 15 | 8.09 (2.18) | 3.21 (2.07) | 3.49 (2.95) | 8.85 (2.83)
  Day 22 | 9.57 (2.90) | 3.6 (2.76) | 3.66 (3.50) | 6.63 (3.36)
  Day 29 | 7.16 (2.41) | 1.53 (2.30) | 4.33 (2.36) | 8.70 (2.26)

4. Secondary Outcome: Moist Wound Environment as Per the Bates-Jensen Wound Assessment Tool (BWAT)
Description: Modified Bates-Jensen Wound Assessment (BWAT-m) Scores for those characteristics measured (wound exudate type and amount) were each graded on a 5-point scale, with 1 being the best and 5 being the worst.
Time Frame: At every visit: Day 8, Day 15, Day 22, Day 29
Measure: Least Squares Mean (Standard Error); unit: BWAT-m Exudate Score
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU
Number analyzed (Participants) | 30 | 33 | 12 | 13
BWAT-m Exudate Score
  Day 8 | 1.94 (0.14) | 1.90 (0.14) | 1.78 (0.20) | 2.43 (0.19)
  Day 15 | 1.78 (0.14) | 1.88 (0.13) | 1.80 (0.25) | 1.95 (0.24)
  Day 22 | 1.76 (0.17) | 1.77 (0.16) | 1.89 (0.32) | 2.24 (0.34)
  Day 29 | 1.69 (0.14) | 1.51 (0.12) | 1.98 (0.37) | 2.02 (0.41)

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | HP828-101 Treating DFU | Standard of Care Treating DFU | HP828-101 Treating PU | Standard of Care Treating PU
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/33 | 0/12 | 1/13
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33 | 0/12 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP828-101 Treating DFU (N=30) | Standard of Care Treating DFU (N=33) | HP828-101 Treating PU (N=12) | Standard of Care Treating PU (N=13)
Infection of ulcer - nontarget ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The severity of the event was Moderate; the Investigator determined that the serious adverse event was not related to the test article. Subject discontinued from the study.
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Study drug dosage was interrupted during the hospitalization. The severity of the event was Moderate; the Investigator determined that the SAE was not related to the test article. Subject discontinued from the study
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The severity of the event was Mild; the Investigator determined that the serious adverse event was not related to the test article. Subject completed the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less